CLINICAL TRIAL: NCT05647382
Title: Soluble Vascular Endothelial-cadherin in Prediction and Diagnosis of Early Postoperative Hypoxemia After Cardiopulmonary Bypass
Brief Title: Soluble VE-cadherin in Prediction and Diagnosis of Early Postoperative Hypoxemia After Cardiopulmonary Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhuan Zhang (Other)
Responsible Party: Sponsor-Investigator, Zhuan Zhang, Director, Yangzhou University
Organization: Yangzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 20221123
Record Dates: First submitted 2022-11-23; First posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Hypoxemia; ARDS; Lung Injury, Acute; Cardiopulmonary Bypass
Keywords: Hypoxemia; acute lung injury; Cardiopulmonary Bypass; FiO2/PaO2
MeSH Terms: conditions — Hypoxia; Acute Lung Injury | interventions — Echocardiography

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lung injury group (Active Comparator): Lung injury is defined as lung damage when the patient has an oxygen and index below 300 24 hours after cardiopulmonary bypass
  Interventions: Diagnostic Test: blood cell analysis, blood gas surveillance, chest radiograph and echocardiography
- Non-lung injury group (Sham Comparator): Patients with oxygen and an index above 300 24 hours after cardiopulmonary bypass are defined as non-lung injury
  Interventions: Diagnostic Test: blood cell analysis, blood gas surveillance, chest radiograph and echocardiography

INTERVENTIONS:
Diagnostic Test: blood cell analysis, blood gas surveillance, chest radiograph and echocardiography — Laboratory parameters of all postoperative patients including blood cell analysis, blood gas surveillance, liver, and kidney function alone with chest radiograph and echocardiography were dynamically monitored.

SUMMARY:
More than 2 million patients worldwide receive heart surgery every year, majority of these surgical patients will undergo cardiopulmonary bypass. However, the incidence of postoperative acute lung injury due to cardiopulmonary bypass is still as high as 20% to 35%. According to clinical experience, the earlier lung damage is detected, the more successful the treatment will be. On the basis of traditional detection, the investigators found a new indicator, serum soluble vascular endothelial-cadherin, which are easy to obtain and have certain specificity. Importantly, they can predict postoperative acute lung injury within 1 hour after cardiac surgery. It is meaningful that this indicator can provide clinicians with early decision-making advice and immediate treatment for patients who may be at risk.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Underwent cardiac surgery using CPB technology.

Exclusion Criteria:

* Patient's lack of consent to participate;
* Presence of abnormal liver, kidney or other organ function;
* Pulmonary inflammation, chronic obstructive pulmonary disease or tumors;
* Underwent cardiac surgery without CPB technology;
* Postoperative need for extracorporeal membrane oxygenation support.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
PaO2/FiO2 ratio | Day 1 after CPB, Day 2 after CPB
  The ratio of inspiratory oxygen fraction to oxygen pressure (PaO2/FiO2) was calculated
lung-injury scores | Day 1 after CPB, Day 2 after CPB
  A structured tutorial was used to establish consensus in the interpretation of radiographs for radiographic lung-injury scores, range from 0 to 4.
  0: No alveolar consolidation; 1: Alveolar consolidation confined to 1 quadrant; 2: Alveolar consolidation confined to 2 quadrants 3: Alveolar consolidation confined to 3 quadrants; 4: Alveolar consolidation in all 4 quadrants.
  The higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Hospital of Yangzhou University, Yangzhou, Jiangsu, China